CLINICAL TRIAL: NCT07012018
Title: Pancreas Screening in High Risk Individuals: A Prospective Cohort
Brief Title: Pancreas Screening in High Risk Individuals
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jennifer Telford, Clinical Professor of Medicine, University of British Columbia
Other Study IDs: H25-01796
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Pancreas Cancer Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High risk individuals for pancreas cancer: Individuals undergoing pancreas screening

SUMMARY:
Pancreas cancer is the 11th most common cancer in Canada but the 4th most common cause of cancer death because by the time pancreas cancer is detected, it is almost always too advanced for surgery. There are known factors that put individuals at higher risk for pancreas cancer. These include: certain genetic mutations, a family history of pancreas cancer, pancreas cysts and a new diagnosis of diabetes mellitus. Individuals with these risk factors are recommended to undergo pancreas screening with blood tests and yearly imaging tests of the pancreas. Our study will enroll patients with these risk factors and ensure they are managed as per guidelines. Prospectively collected data will include: patient clinicodemographic details, lifestyle factors, screening test results, clinical outcomes and patient reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Family history of pancreatic cancer, pathogenic variant increasing risk of pancreatic cancer, IPMN, new onset diabetes.

Exclusion Criteria:

* Unable to give informed consnet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High risk individuals referred for pancreas screening
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of pancreatic cancer | 10 years

IPD SHARING:
Plan to Share IPD: No